CLINICAL TRIAL: NCT01657578
Title: Optimal Dose and Population Pharmacokinetics of Omeprazole in Neonates With Gastroesophageal Reflux Disease (GERD)
Brief Title: Optimal Dosing of Omeprazole in Neonates
Acronym: OMEPRAZOLE-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P 051043; 2006-005335-16 (EudraCT Number)
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-07

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: neonates; reflux disease; population pharmacokinetics, omeprazole
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- neonates of less than 32 weeks gestational age (Experimental): omeprazole
  Interventions: Drug: Omeprazole
- neonates born between 32 and 35 weeks of GA (Experimental): omeprazole
  Interventions: Drug: Omeprazole
- neonates of more than 36 weeks of GA (Experimental): omeprazole
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole — administration of Omeprazole
  Other Names: administration of Omeprazole

SUMMARY:
"The principal aim of this trial is to determine the minimum effective dose of omeprazole in neonates with GERD objectively diagnosed by a 24-h intra-oesophageal pH monitoring (pHmetry), to obtain a short-term efficacy in the pHmetry of control performed 72 hrs ± 24 after initiation of omeprazole.

The secondary objectives of the study were: (1) to assess the efficacy of omeprazole upon other pHmetry parameters, (2) to characterize the population pharmacokinetics and pharmacogenetics of omeprazole, (3) to evaluate the effect of omeprazole upon oro-pharyngeal pH monitoring and (4) to assess the short-term safety of use of omeprazole in neonates."

DETAILED DESCRIPTION:
"Omeprazole is a proton pump inhibitor increasingly prescribed in the neonatal population for gastroesophageal reflux disease (GERD) complicated or not by the presence of esophagitis. Although extensively evaluated in adults, optimal dosing schemas, efficacy and safety have not been determined in the neonatal population where its prescription remains off-label. The study is a double blind trial that was designed using a Bayesian sequential analysis approach. The principle of this approach is to identify the adequate drug dosage to obtain a level of efficacy as close as possible to a predetermined target level of efficacy in the population. In this study, five different dosages of omeprazole are tested (1, 1,5, 2, 2,5, 3 mg/kg/day) and a target probability of successful treatment of 95% has been chosen. To assess the influence of gestational age on omeprazole's efficacy, analysis was stratified on 3 groups: (1) neonates of less than 32 weeks gestational age (GA), (2) neonates born between 32 and 35 weeks of GA, (3) neonates of more than 36 weeks of GA.

A total maximum number of 90 neonates is expected to be included (30 neonates per group).

Patients' participation in the study ends after completion of the pHmetry of control that is 72 ±24 hours after omeprazole initiation.

Patients in the study will all benefit for the management of their GERD from non-pharmacological therapies such as adequate positioning and use of available thickening agents for formula The only pharmacologic agent authorised during study for treating GERD is omeprazole. All other available GERD treatments will not be prescribed."

ELIGIBILITY:
INCLUSION CRITERIA:

* Full-term neonates or preterm neonates with a postmenstrual age >/= 35 weeks
* Presenting abnormal pHmetry (= percentage of the entire record that intra-oesophageal pH is <4 is superior or equal to 5%)
* Patient must receive discontinuous oral feedings
* If proton pump inhibitors or other pharmacologic antireflux therapies had already commenced, these had to be withdrawn 7 days before baseline recordings
* In-patient in Neonatal Intensive Care Unit or Neonatology Unit of the Robert Debré University Hospital
* Both parents sign written informed consent form
* Affiliated to social security

EXCLUSION CRITERIA:

* Patients under proton pump inhibitors (PPI) treatment or that have discontinued PPI treatment less than 7 days before inclusion
* Patients with acute gastrointestinal disease (diarrhoea)
* Patients than present leucopenia or thrombocytopenia (value half the normal value for age)
* Patients that present aspartate and alanine aminotransferase values twice the upper limit of normal
* Patients that present renal and hepatic failure
* Newborns presenting galactosemia, glucose-galactose malabsorption, deficiency in lactase enzymes
* Co-administration of atazanavir and ritonavir
* Patients allergic to omeprazole or to any other ingredients in the medicine

Min Age: 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-06; Primary Completion 2010-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Presence of a normalised control pHmetry Presence of a normalised control pHmetry Presence of a normalised control pHmetry | 72±24 hours after initiation of omeprazole treatment
  Normalised control pHmetry is defined by a reflux index (duration that the recorded intra-oesophageal pH is less than 4.0, expressed as a percentage of the total duration of pH monitoring) of less than 5%

SECONDARY OUTCOMES:
mean number of reflux episodes per hour | 72±24 hours after initiation of omeprazole treatment
  mean number of reflux episodes per hour
duration of the longest reflux episode | 72±24 hours after initiation of omeprazole treatment
  duration of the longest reflux episode
plasma concentrations of omeprazole and its metabolite, hydroxyl-omeprazole | H0.5 and H4 or between H4 and H12 after the first administration of omeprazole
  Plasma concentrations of omeprazole and its metabolite, hydroxyl-omeprazole, After the first administration of omeprazole, blood will be collected either between H0.5 and H4 or between H4 and H12 or both
changes in salivary pH monitoring | just before and 3 hours after a meal Under treatment period
  changes in salivary pH monitoring Without treatment period: just before and 3 hours after a meal Under treatment period: just before and just after the insertion of the pHmetry catheter
changes in biological parameters | 96±24 hours after initiation of omeprazole treatment
  changes in biological parameters

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne Jacqz-Aigrain, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hospital Robert Debre, Paris, France